CLINICAL TRIAL: NCT05145283
Title: Recombinant Human C1 Esterase Inhibitor (Conestat Alfa) in the Prevention of Acute Ischemic Cerebral and Renal Events After Transcatheter Aortic Valve Implantation: a Multi-center, Randomized, Double-blind, Placebo-controlled Investigational Study (PAIR-TAVI).
Brief Title: Recombinant Human C1 Esterase Inhibitor (Conestat Alfa) in the Prevention of Acute Ischemic Cerebral and Renal Events After Transcatheter Aortic Valve Implantation
Acronym: PAIR-TAVI
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Swiss National Science Foundation (Other); Pharming Technologies B.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2021-02025; me19Osthoff
Record Dates: First submitted 2021-11-17; First posted 2021-12-06 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Acute Ischemic Stroke; Acute Renal Injury
Keywords: Severe aortic stenosis (AS); Valvular heart disease; Transcatheter aortic valve implantation (TAVI); cerebral embolic events; renal embolic events; Ischemia/reperfusion injury (IRI); recombinant human C1 esterase inhibitor (rhC1INH, conestat alfa); complement system; contact activation system
MeSH Terms: conditions — Ischemic Stroke; Acute Kidney Injury; Aortic Valve Stenosis; Heart Valve Diseases; Reperfusion Injury | interventions — conestat alfa; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Patients will be randomized in two parallel groups to receive either conestat alfa or placebo.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conestat alfa (Ruconest®) intervention group (Active Comparator): The intervention group will receive conestat alfa (Ruconest®) as a 10-minute slow intravenous injection (up to 56 ml) once during the TAVI procedure followed by a second administration (up to 28 ml) again three hours later. The first administration will include a dosage of 100 U/kg (maximum 8400 U) conestat alfa. The dosing of the second administration will be 50 U/kg (maximum 4200 U).
  Interventions: Drug: Conestat alfa (Ruconest®)
- saline injection placebo group (Placebo Comparator): Subjects randomized into the placebo group will receive an intravenous normal saline injection with corresponding volume over 10 minutes during the TAVI procedure and three hours later after the first administration.
  Interventions: Drug: NaCl 0.9%)

INTERVENTIONS:
Drug: Conestat alfa (Ruconest®) — In the current study, participants will receive two intravenous injections of conestat alfa (immediately during the TAVI procedure and again 3h later) at a dose of 100 U/kg (first dose) and of 50 U/kg (subsequent dose), for patients less than 84 kg; two intravenous injections (immediately during the TAVI procedure and again 4h later) of conestat at a dose of 8400 U (4 vials, first dose) and of 4200 U (2 vials, subsequent dose) for patients of 84 kg body weight or greater. The chosen regimen including repeated administration should increase and maintain serum C1INH levels above twice the serum concentration for six to eight hours in the majority of patients. The timeframe of therapeutic concentrations will cover the period of the TAVI procedure itself and the immediate postprocedural period during which reperfusion and additional ischemic events related to global hypoperfusion may occur.
  Arms: Conestat alfa (Ruconest®) intervention group
Drug: NaCl 0.9%) — Normal saline (NaCl 0.9%) will serve as placebo treatment. The respective amount of saline (according to patient weight matching the volume of conestat alfa that would have been used for this patient) will be withdrawn in an opaque syringe for slow IV injection.
  Arms: saline injection placebo group

SUMMARY:
The aim of this trial is to assess the safety and efficacy of conestat alfa (Ruconest®, Pharming Technologies B.V.) on renal and cerebral ischemic events in patients undergoing TAVI for severe symptomatic aortic stenosis (AS) compared to placebo.

DETAILED DESCRIPTION:
Severe aortic stenosis (AS) is a frequent valvular heart disease in the elderly with a prevalence of 4 to 10% and a mean survival of only 0.5 to 5 years if left untreated. Transcatheter aortic valve implantation (TAVI) has evolved as standard of care for high-, intermediate and potentially even low surgical risk candidates due to a lower perioperative risk compared to surgical aortic valve replacement (SAVR). Despite its relative safety compared to SAVR, embolic events originating from the calcified valve and leading to ischemic stroke and acute renal injury are major complications following TAVI in the acute and subacute period, and are associated with increased morbidity including cognitive decline and mortality. While cerebral embolic protection devices (CEPD) such as the Sentinel® CEPD (Boston Scientific) were designed to reduce the burden of cerebral embolic events, their impact on clinical events has yet to be determined, and other prophylactic options are currently not available. Ischemia/reperfusion injury (IRI) is a key pathophysiological mechanism involved in cerebral and renal embolic events after TAVI resulting in activation of endothelial cells, the contact activation and the complement system and attraction of neutrophils to the site of injury. In this regard, recombinant human C1 esterase inhibitor (rhC1INH, conestat alfa), a potent inhibitor of the complement and the contact system has been shown to reduce the size of cerebral ischemic damage and of renal injury in experimental IRI models, and has successfully been investigated in a pilot study of acute kidney injury following the administration of contrast media. The aim of the current trial is to assess the safety and efficacy of conestat alfa (Ruconest®, Pharming Technologies B.V.) on renal and cerebral ischemic events in patients undergoing TAVI for severe symptomatic AS compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent as documented by signature
* Severe AS and scheduled for transfemoral TAVI

Exclusion Criteria:

* Contraindications to the class of drugs under study (C1INH), e.g., known hypersensitivity or allergy to class of drugs or the investigational product
* History of allergy to rabbits (as rhC1INH is derived from the breast milk of transgenic rabbits)
* Women who are pregnant or breast feeding
* Hemodynamic instability requiring emergency TAVI
* Valve-in-valve procedure
* Other access route than transfemoral
* Non-cardiac co-morbidity with expected survival <6 months
* Ischemic or hemorrhagic stroke within 30 days before TAVI
* Dialysis or estimated glomerular filtration rate (eGFR) <20 ml/min/1.73m2
* Contraindication for MRI such as a permanent non-MRI compatible pacemaker or severe claustrophobia
* Liver cirrhosis (any Child-Pugh score)
* Incapacity or inability to provide informed consent
* Participation in another study with investigational drug or medical device within the 30 days preceding and during the present study
* Previous enrolment into the current study
* Any uncontrolled or significant concurrent illness that would put the patient at a greater risk or limit compliance with the study requirements at the discretion of the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2022-03-16 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Total volume of new cerebral ischemic lesions as evaluated by magnetic resonance imaging (MRI) | on day 4 (+/-1 day) after transfemoral TAVI
  Total volume of new cerebral ischemic lesions as evaluated by magnetic resonance imaging (MRI)

SECONDARY OUTCOMES:
Maximum new lesion volume as measured by MRI (i.e. volume of the largest new lesion) | on day 4 (+/-1 day) after transfemoral TAVI
  Maximum new lesion volume as measured by MRI (i.e. volume of the largest new lesion)
Number of new cerebral ischemic lesions as measured by MRI | on day 4 (+/-1 day) after transfemoral TAVI
  Number of new cerebral ischemic lesions as measured by MRI
Number (incidence) of clinically manifest ischemic stroke | within 48 hours after TAVI
  Number (incidence) of clinically manifest ischemic stroke
Change in secondary brain atrophy at 3-months follow-up | at baseline and at 3-months follow-up
  Secondary brain atrophy at 3-months follow-up related to the gradual cellular loss as measured by high resolution 3D T1-weighted MR images (defined as the difference between the brain volumes)
Change in secondary infarct growth at 3-months follow-up (defined as the difference between the infarct volumes) | at day 4 and at 3-months
  Change in secondary infarct growth at 3-months follow-up (defined as the difference between the infarct volumes)
Total brain damage (defined as the sum of secondary brain atrophy and final infarct volume) | at 3 months
  Total brain damage (defined as the sum of secondary brain atrophy and final infarct volume)
Change in National Institutes of Health Stroke Scale Score (NIHSS) | at baseline and at 3-months follow-up
  The NIHSS is composed of 11 items, each of which scores a specific ability between a 0 and 4. For each item, a score of 0 typically indicates normal function in that specific ability, while a higher score is indicative of some level of impairment. The individual scores from each item are summed in order to calculate a patient's total NIHSS score. The maximum possible score is 42, with the minimum score being a 0.
Change in modified Rankin scale | at baseline and at 3-months follow-up
  Change in modified Rankin scale; scale runs from 0-6, running from perfect health (0) without symptoms to death (6)
Change in trail making test | at baseline and at 3-months follow-up
  Change in trail making test; scoring is based on time taken to complete the test (e.g. 35 seconds yielding a score of 35) with lower scores being better.
Change in Montreal Cognitive Assessment test (MOCA) | at baseline and at 3-months follow-up
  Montreal Cognitive Assessment test scores range between 0 and 30. A score of 26 or over is considered to be normal
Incidence of acute kidney injury (AKI) defined according to the Kidney Disease: Improving Global Outcomes criteria (any stage) | within 3 days after TAVI
  Incidence of AKI defined according to the Kidney Disease: Improving Global Outcomes criteria (any stage)
Peak increase of urinary Neutrophil Gelatinase-Associated Lipocalin (NGAL) | within 48 hours after TAVI
  Peak increase of urinary NGAL (surrogate marker of acute renal injury)
Incidence of significant increase in serum cystatin C (>10%) | within 48 hours after TAVI
  Incidence of significant increase in serum cystatin C (>10%)

OTHER OUTCOMES:
Persistent renal impairment after 3 months (defined as increase in serum creatinine of at least 50% from baseline at 3 months) | at 3-months follow-up
  Persistent renal impairment after 3 months (defined as serum creatinine increase of at least 50% from baseline at 3 months)
Change in concentration of C1-Esterase-Inhibitor (C1INH) | during the first 24 hours after TAVI
  Change in concentration of C1INH
Change in troponin T to assess myocardial injury following TAVI | within 72 hours after TAVI
  Change in troponin T to assess myocardial injury following TAVI
Change in urinary biomarkers of renal injury (Kidney Injury Molecule-1 (KIM-1) and osteopontin) | within 48 hours after TAVI
  Change in urinary biomarkers of renal injury (Kidney Injury Molecule-1 (KIM-1) and osteopontin)
Change in serum neurofilament light chain (marker of neuroaxonal damage) | within 3 months after TAVI
  Change in serum neurofilament light chain (marker of neuroaxonal damage)
Number of adverse events | within 3 months after TAVI
  Number of adverse events
Number of serious adverse events | within 3 months after TAVI
  Number of serious adverse events
Number of major cardiovascular and renal events (cardiovascular death, non-fatal myocardial infarction, heart failure hospitalization, stroke, dialysis) | within 3 months after TAVI
  Number of major cardiovascular and renal events (cardiovascular death, non-fatal myocardial infarction, heart failure hospitalization, stroke, dialysis)
Number of complications of transfemoral TAVI | within 3 months after TAVI
  Number of complications of transfemoral TAVI such as conduction disturbance (including permanent pacemaker implantation) or aortic regurgitation according to the Valve Academic Research Consortium (VARC)-3 criteria, or bleeding according to the Bleeding Academic Research Consortium (BARC)-criteria)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Osthoff, Prof. Dr. med., Principal Investigator — University Hospital Basel, Division of Internal Medicine; Raban Jeger, Prof. Dr. med., Principal Investigator — Stadtspital Triemli Zürich, Division of Cardiology
Locations (2):
- Switzerland (2):
  - University Hospital Basel, Division of Internal Medicine, Basel
  - Stadtspital Triemli Zürich, Division of Cardiology, Zurich